CLINICAL TRIAL: NCT02970318
Title: A Randomized, Multicenter, Open-Label, Phase 3 Study of Acalabrutinib (ACP-196) Versus Investigator's Choice of Either Idelalisib Plus Rituximab or Bendamustine Plus Rituximab in Subjects With R/R Chronic Lymphocytic Leukemia
Brief Title: A Study of Acalabrutinib vs Investigator's Choice of Idelalisib Plus Rituximab or Bendamustine Plus Rituximab in R/R CLL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACE-CL-309; 2015-004454-17 (EudraCT Number)
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; BTK; Bruton Tyrosine Kinase; acalabrutinib; ACP-196
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; Rituximab; idelalisib; Bendamustine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acalabrutinib (ACP-196) (Experimental): Acalabrutinib (ACP-196) Monotherapy
  Interventions: Drug: Acalabrutinib (ACP-196)
- Rituximab Plus Idelalisib or Bendamustine (Active Comparator): Investigator's Choice of Rituximab Plus Idelalisib or Bendamustine
  Interventions: Drug: Rituximab; Drug: Idelalisib; Drug: Bendamustine

INTERVENTIONS:
Drug: Acalabrutinib (ACP-196) — Acalabrutinib monotherapy
  Arms: Acalabrutinib (ACP-196)
Drug: Rituximab — Rituximab in combination with idelalisib or bendamustine
  Arms: Rituximab Plus Idelalisib or Bendamustine
Drug: Idelalisib — Idelalisib in combination with rituximab
  Arms: Rituximab Plus Idelalisib or Bendamustine
Drug: Bendamustine — Bendamustine in combination with rituximab
  Arms: Rituximab Plus Idelalisib or Bendamustine

SUMMARY:
This study is designed to evaluate the efficacy of acalabrutinib compared with rituximab in combination with idelalisib or bendamustine in previously treated subjects with chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. ECOG performance status of 0 to 2.
3. Diagnosis of CLL that meets published diagnostic criteria (Hallek 2008):

   1. Monoclonal B-cells (either kappa or lambda light chain restricted) that are clonally co-expressing ≥ 1 B-cell marker (CD19, CD20, or CD23) and CD5.
   2. Prolymphocytes may comprise ≤ 55% of blood lymphocytes.
   3. Presence of ≥ 5 x 10^9 B lymphocytes/L (5000/μL) in the peripheral blood (at any point since initial diagnosis).
4. Must have documented CD20-positive CLL.
5. Active disease meeting ≥ 1 of the following IWCLL 2008 criteria for requiring treatment:

   1. Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia (hemoglobin < 10 g/dL) and/or thrombocytopenia (platelets < 100,000/μL).
   2. Massive (i.e., ≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
   3. Massive nodes (i.e., ≥ 10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy.
   4. Progressive lymphocytosis with an increase of > 50% over a 2-month period or a LDT of < 6 months. LDT may be obtained by linear regression extrapolation of ALC obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In subjects with initial blood lymphocyte counts of < 30 x 10^9/L (30,000/μL), LDT should not be used as a single parameter to define indication for treatment. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (e.g., infections) should be excluded.
   5. Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy.
   6. Constitutional symptoms documented in the subject's chart with supportive objective measures, as appropriate, defined as ≥ 1 of the following disease-related symptoms or signs:

   i. Unintentional weight loss ≥ 10% within the previous 6 months before screening.

   ii. Significant fatigue (ECOG performance score 2; inability to work or perform usual activities).

   iii. Fevers higher than 100.5°F or 38.0°C for ≥ 2 weeks before screening without evidence of infection.

   iv. Night sweats for > 1 month before screening without evidence of infection.
6. Meet the following laboratory parameters:

   1. ANC ≥ 750 cells/μL (0.75 x 10^9/L), or ≥ 500 cells/μL (0.50 x 10^9/L) in subjects with documented bone marrow involvement, and independent of growth factor support 7 days before assessment.
   2. Platelet count ≥ 50,000 cells/μL (50 x 10^9/L), or ≥ 30,000 cells/μL (30 x 10^9/L) in subjects with documented bone marrow involvement, and without transfusion support 7 days before assessment. Subjects with transfusion-dependent thrombocytopenia are excluded. If an Investigator has chosen bendamustine/rituximab as the Arm B treatment, platelets must be ≥ 75,000 cells/μL (75 x 10^9/L).
   3. Serum AST and ALT ≤ 2.0 x ULN.
   4. Total bilirubin ≤ 1.5 x ULN.
   5. Estimated creatinine clearance of ≥ 30 mL/min, calculated using the formula of Cockcroft and Gault [(140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female].
7. Must have received ≥ 1 prior systemic therapies for CLL. Note: Single-agent steroids or localized radiation are not considered a prior line of therapy. If a single-agent anti-CD20 antibody was previously administered, subjects must have received ≥ 2 doses.
8. Women who are sexually active and can bear children must agree to use highly effective forms of contraception while on the study and for 2 days after the last dose of acalabrutinib, 90 days after the last dose of idelalisib, 6 months after the last dose of bendamustine, or 12 months after the last dose of rituximab, whichever is longer. Highly effective forms of contraception are defined in Section 9.2.5.
9. Men who are sexually active and can beget children must agree to use highly effective forms of contraception during the study and for 90 days after the last dose of idelalisib, 6 months after the last dose of bendamustine, or 12 months after the last dose of rituximab, whichever is longer. Highly effective forms of contraception are defined in Section 9.2.5.
10. Men must agree to refrain from sperm donation during the study and for 90 days after the last dose of idelalisib, 6 months after the last dose of bendamustine, or 12 months after the last dose of rituximab, whichever is longer.
11. Willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules without difficulty.
12. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Exclusion Criteria:

1. Known CNS lymphoma or leukemia.
2. Known prolymphocytic leukemia or history of, or currently suspected, Richter's syndrome.
3. Uncontrolled AIHA or ITP defined as declining hemoglobin or platelet count secondary to autoimmune destruction within the screening period or requirement for high doses of steroids (> 20 mg daily of prednisone or equivalent).
4. Prior exposure to a BCL-2 inhibitor (e.g., venetoclax/ABT-199) or a BCR inhibitor (e.g., BTK inhibitors or PI3K inhibitors). Prior bendamustine is allowed if Investigator's choice for treatment in Arm B is idelalisib with rituximab. Bendamustine retreatment is allowed if the prior response to bendamustine lasted > 24 months.
5. Received any chemotherapy, external beam radiation therapy, anticancer antibodies, or investigational drug within 30 days before first dose of study drug.
6. Corticosteroid use > 20 mg daily prednisone equivalent within 1 week before first dose of study drug, except as indicated for other medical conditions such as inhaled steroid for asthma, topical steroid use, or as premedication for administration of study drug or contrast. For example, subjects requiring steroids at daily doses > 20 mg prednisone equivalent systemic exposure daily, or those who are administered steroids for leukemia control or white blood cell count lowering are excluded.
7. Prior radio- or toxin-conjugated antibody therapy.
8. Prior allogeneic stem cell transplant or prior autologous transplant within 6 months of first dose of study drug(s) or presence of graft-vs-host disease or receiving treatment for graft-vs-host disease.
9. Major surgical procedure within 30 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
10. History of prior malignancy except for the following:

    1. Malignancy treated with curative intent and with no evidence of active disease present for more than 2 years before screening and felt to be at low risk for recurrence by treating physician.
    2. Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled nonmelanomatous skin cancer.
    3. Adequately treated carcinoma in situ without current evidence of disease.
11. Significant cardiovascular disease such as uncontrolled or untreated symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or QTc > 480 msec (calculated using Fridericia's formula: QT/RR^0.33) at screening. Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll on study.
12. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach, or extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
13. Received a live virus vaccination within 28 days of first dose of study drug.
14. Known history of infection with HIV or any uncontrolled active systemic infection (e.g., bacterial, viral, or fungal). For study sites in Germany: active infection with human immunodeficiency virus (seropositivity for HIV-1 or HIV-2 antibodies, and if positive, reactivity against the HIV-specific p24 antigen).
15. Active CMV infection (active viremia as evidenced by positive polymerase chain reaction [PCR] result for CMV DNA).
16. Serologic status reflecting active hepatitis B or C infection.

    1. Subjects who are anti-HBc positive and who are surface antigen negative will need to have a negative PCR result before randomization. Those who are HbsAg-positive or hepatitis B PCR positive will be excluded.
    2. Subjects who are hepatitis C antibody positive will need to have a negative PCR result before randomization. Those who are hepatitis C PCR positive will be excluded.
17. Ongoing, drug-induced liver injury, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
18. History of or ongoing drug-induced pneumonitis.
19. History of serious allergic reactions including anaphylaxis and toxic epidermal necrolysis.
20. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
21. History of bleeding diathesis (e.g., hemophilia, von Willebrand disease).
22. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of first dose of study drug.
23. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
24. Requires treatment with a strong CYP3A inhibitor/inducer.
25. Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
26. Breast feeding or pregnant.
27. Concurrent participation in another therapeutic clinical trial.
28. Prothrombin time/INR or aPTT (in the absence of a Lupus anticoagulant) > 2.0 x ULN. Exception: Subjects receiving warfarin are excluded, however, those receiving other anticoagulant therapy who have a higher INR/aPTT may be permitted to enroll to this study after discussion with the medical monitor.
29. History of confirmed progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2027-10-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (143):
- United States (13):
  - Research Site, Chandler, Arizona
  - Research Site, Oxnard, California
  - Research Site, Athens, Georgia
  - Research Site, Joliet, Illinois
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Mount Sterling, Kentucky
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Brick, New Jersey
  - Research Site, Nyack, New York
  - Research Site, Canton, Ohio
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Round Rock, Texas
- Australia (11):
  - Research Site, Adelaide
  - Research Site, Box Hill
  - Research Site, Frankston
  - Research Site, Geelong
  - Research Site, Gosford
  - Research Site, Hobart
  - Research Site, Kogarah
  - Research Site, Murdoch
  - Research Site, Nedlands
  - Research Site, South Brisbane
  - Research Site, Woodville
- Austria (4):
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (4):
  - Research Site, Antwerp
  - Research Site, Ghent
  - Research Site, Roeselare
  - Research Site, Yvoir
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Stara Zagora
  - Research Site, Vratsa
- Canada (7):
  - Research Site, Barrie, Ontario
  - Research Site, Calgary
  - Research Site, Montreal
  - Research Site, Ottawa
  - Research Site, Regina
  - Research Site, Saint John
  - Research Site, Toronto
- Croatia (2):
  - Research Site, Zadar
  - Research Site, Zagreb
- Czechia (6):
  - Research Site, Brno
  - Research Site, Nový Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava Poruba
  - Research Site, Plzen - Lochotin
  - Research Site, Prague
- France (9):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Provence Alpes Cote D'Azur
  - Research Site, Rennes
  - Research Site, Rouen
- Germany (5):
  - Research Site, Aschaffenburg
  - Research Site, Dresden
  - Research Site, Mutlangen
  - Research Site, München
  - Research Site, Ulm
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Pok Fu Lam
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Kaposvár
- Israel (6):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Petah Tikvah
- Italy (8):
  - Research Site, Aviano
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
- New Zealand (4):
  - Research Site, Addington
  - Research Site, Dunedin
  - Research Site, Palmerston North
  - Research Site, Tauranga
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Woj. Podkarpackie
- Russia (10):
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Penza
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Sochi
  - Research Site, Tula
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Research Site, SGP, Singapore
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Košice
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Donggu
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seoul
- Spain (6):
  - Research Site, Badalona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Salamanca
  - Research Site, Santander
  - Research Site, Valencia
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Luleå
  - Research Site, Stockholm
- Taiwan (3):
  - Research Site, Hualien City
  - Research Site, Tainan
  - Research Site, Taipei
- Ukraine (6):
  - Research Site, Cherkasy
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Khmelnytsky
  - Research Site, Kyiv
  - Research Site, Zhytomyr
- United Kingdom (9):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Canterbury
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Manchester
  - Research Site, Southampton
  - Research Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Eek D, Ivanescu C, Corredoira L, Meyers O, Cella D. Content validity and psychometric evaluation of the Functional Assessment of Chronic Illness Therapy-Fatigue scale in patients with chronic lymphocytic leukemia. J Patient Rep Outcomes. 2021 Mar 11;5(1):27. doi: 10.1186/s41687-021-00294-1. PMID 33709202
- [Derived] Ghia P, Pluta A, Wach M, Lysak D, Kozak T, Simkovic M, Kaplan P, Kraychok I, Illes A, de la Serna J, Dolan S, Campbell P, Musuraca G, Jacob A, Avery E, Lee JH, Liang W, Patel P, Quah C, Jurczak W. ASCEND: Phase III, Randomized Trial of Acalabrutinib Versus Idelalisib Plus Rituximab or Bendamustine Plus Rituximab in Relapsed or Refractory Chronic Lymphocytic Leukemia. J Clin Oncol. 2020 Sep 1;38(25):2849-2861. doi: 10.1200/JCO.19.03355. Epub 2020 May 27. PMID 32459600
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-309&attachmentIdentifier=4d2fac79-d899-4138-8657-0bb2b540784b&fileName=ace-cl-309-csp-amend-8-redact.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-309&attachmentIdentifier=5ba8b7a4-ac40-4f7a-b333-9c025218e080&fileName=ace-cl-309-sap-ed-3-redact.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-309&attachmentIdentifier=aa63aaa7-e136-4da4-89c9-2ad21beb4457&fileName=ace-cl-309-Study_Synopsis-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Randomized, Multicenter, Open-Label, Phase 3 Study of Acalabrutinib (ACP-196) Versus Investigator's Choice of Either Idelalisib Plus Rituximab or Bendamustine Plus Rituximab in Subjects with Relapsed or Refractory Chronic Lymphocytic Leukemia. A total of 310 subjects met the eligibility criteria and were randomized to the acalabrutinib arm (N = 155) and IR/BR arm (N = 155).
  All but 3 subjects (1 randomized to acalabrutinib and 2 randomized to IR/BR) received study treatment.
Pre-assignment Details: 310 patients were enrolled in this study and agreed to move forward in participating in the trial.
Groups:
- Arm A- Acala 100 mg BID- Overall Study Period: Arm A- Acalabrutinib 100 mg BID- Overall Study Period
- Arm B: Investigator Choice (IR or BR)-Main Study Period: IR or BR data not presented separately similar to combined treatment arms approved for D8223C00009
- Arm B- Inv Choice of IR Crossed Over to Arm A- Acala. 100 mg BID: Arm B- Investigator Choice of IR Crossed Over to Arm A- Acala. 100 mg BID
- Arm B- Inv. Choice of BR Crossed Over to Arm A- Acala. 100 mg BID: Arm B- Investigator Choice of BR Crossed Over to Arm A- Acala. 100 mg BID
Period: Overall for Arm A & Main for Arm B
Arm/Group | Arm A- Acala 100 mg BID- Overall Study Period | Arm B: Investigator Choice (IR or BR)-Main Study Period | Arm B- Inv Choice of IR Crossed Over to Arm A- Acala. 100 mg BID | Arm B- Inv. Choice of BR Crossed Over to Arm A- Acala. 100 mg BID
Started | 155 | 155 | 0 | 0
Arm B Treatment= Idelalisib Plus Rituximab | 0 | 119 | 0 | 0
Arm B Treatment = Bendamustine Plus Rituximab | 0 | 36 | 0 | 0
Completed (Completed study treatment at final DCO (03Sep2021)) | 0 | 1 (This subject received 1st dose of study drug on 11Nov2011, completed study treatment on 14MAR2019, never crossed over, and and died 11 months after completing study treatment on 15Feb2020.) | 0 | 0
Completed (Patients ongoing treatment at final DCO (03Sep2021)) | 99 | 26 | 0 | 0
Completed (Patients Ongoing Treatment + Patients Completed Study Treatment at Final DCO (03Sep2021)) | 99 (All 99 subjects ongoing treatment at final DCO.) | 27 (26 subjects ongoing treatment + 1 subject completed study treatment and died 11 months after completing study treatment on 15Feb2020.) | 0 | 0
Not Completed | 56 | 128 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 14 | 0 | 0
Not completed — Death | 41 | 33 | 0 | 0
Not completed — Arm B Crossed Over to Arm A Acala 100 mg Monotherapy | 0 | 80 | 0 | 0
Period: ArmB: Inv.Choice Crossed Over to Acala
Arm/Group | Arm A- Acala 100 mg BID- Overall Study Period | Arm B: Investigator Choice (IR or BR)-Main Study Period | Arm B- Inv Choice of IR Crossed Over to Arm A- Acala. 100 mg BID | Arm B- Inv. Choice of BR Crossed Over to Arm A- Acala. 100 mg BID
Started | 0 | 0 (N/A. Note: No subjects stayed in Arm: Investigator's choice of IR/BR during cross-over period.) | 63 (Note: There were a total of 80 subjects in Arm B crossing over to Arm A shown under the last row of Main Study Period. Among them 63 were randomized to Arm B: IR and 17 were randomized to BR.) | 17 (Note: There were a total of 80 subjects in Arm B crossing over to Arm A shown under the last row of Main Study Period. Among them 63 were randomized to Arm B: IR and 17 were randomized to BR.)
Completed (Ongoing Treatment at Final DCO (03Sep2021)) | 0 | 0 | 42 | 14
Not Completed | 0 | 0 | 21 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 18 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-Treat (ITT) population, which included all randomized participants grouped according to assigned treatment.
Groups:
- Arm A- Acala. 100 mg BID: Arm A- Acalabrutinib 100 mg BID
- Total: Total of all reporting groups
Arm/Group | Arm A- Acala. 100 mg BID | Arm B: Investigator Choice (IR or BR)-Main Study Period | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Customized [Number; unit: Participants]
  Age < 65 Years | 58 | 57 | 115
  Age >=65 years | 97 | 98 | 195
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 55 | 102
  Male | 108 | 100 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 147 | 129 | 276
  Unknown or Not Reported | 6 | 20 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 145 | 141 | 286
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: Participants]
  North America | 8 | 9 | 17
  Australia | 6 | 6 | 12
  New Zealand | 3 | 1 | 4
  Europe | 131 | 132 | 263
  Taiwan, Province Of China | 1 | 0 | 1
  Hong Kong | 0 | 1 | 1
  Korea, Republic Of | 3 | 4 | 7
  Singapore | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Independent Review Committee (IRC) Assessment
Description: To evaluate the efficacy of acalabrutinib monotherapy (Arm A) compared with idelalisib/rituximab or bendamustine/rituximab (Arm B) based on Independent Review Committee (IRC) assessment of progression-free survival (PFS) per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria (Hallek 2008) with incorporation of the clarification for treatment-related lymphocytosis (Cheson 2012) hereafter referred to as IWCLL 2008 criteria in subjects with relapsed or refractory (R/R) chronic lymphocytic leukemia (CLL). As planned and reported in the interim clinical study report (dated 17 July 2019), because the study did cross the boundary at interim analysis.
  IRC assessments were discontinued after the interim analysis. All IRC-related efficacy analyses in this clinical study report were based on the interim analysis data cutoff date of 15 January 2019. All other efficacy analyses were based on the final analysis data cutoff date of 03 September 2021.
Time Frame: IRC assessments from randomization date until disease progression or death or IRC discontinuation on 15Jan2019 (as IA per this data cutoff showed crossing superiority boundary) whichever came first, up to 22 months of follow-up
Population: Intent-to-treat population including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A: Acalabrutinib Monotherapy: Acalabrutinib 100 mg orally twice a day
- Arm B: Investigators Choice: Idelalisib+Rituximab or Bendamustine + Retuximab
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigators Choice
Number analyzed (Participants) | 155 | 155
Months | NA [NA to NA] — Kaplan-Meier Estimated Median PFS and 95% were not reached for Arm A. | 16.5 [14.0 to 17.1]
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigators Choice; Test type: Other; p < 0.0001, Log Rank — Stratified by randomization stratification factors as recorded in IXRS, i.e., presence of del17p (Yes/No), ECOG (0-1/2), # of prior therapies (1-3/4+); Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.20 to 0.49] — Cox Proportional Hazard Model (Arm A vs. Arm B) stratified by factors as recorded in IXRS, i.e., presence of del17p (Yes/No), ECOG (0-1/2), # of prior therapies (1-3/4+)

2. Secondary Outcome: Progression-free Survival (PFS) Per Investigator Assessment
Description: PFS per investigator assessment based on the final analysis data cutoff date of 03 September 2021.
Time Frame: From randomization date to date of disease progression or death due to any cause or data cutoff date on 03Sep2021, whichever came first, regardless of use of subsequent anticancer therapy, until 53 months of follow-up.
Population: Intent-to-treat population including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm B: Investigator's Choice: Idelalisib+Rituximab or Bendamustine + Retuximab
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigator's Choice
Number analyzed (Participants) | 155 | 155
Months | NA [45.8 to NA] — Kaplan-Meier Estimates for median PFS and upper 95% CI were not reached for Arm A. | 16.8 [14.1 to 22.5]
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigator's Choice; Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.20 to 0.38] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: IRC-assessed Overall Response Rate (ORR) Per IWCLL 2008 Criteria Based on Data Cutoff 15 January 2019 From Interim Analysis
Description: IRC-assessed overall response rate (ORR) including complete response (CR), CR with incomplete blood count recovery (CRi) nodular PR (nPR), and Partial Response (PR)
Time Frame: as for outcome 1
Population: Intent-to-treat population including all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigator's Choice
Number analyzed (Participants) | 155 | 155
Participants | 126 | 117
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigator's Choice; Test type: Other; p = 0.2248, Cochran-Mantel-Haenszel; Based on Cochran-Mantel-Haenszel test with adjustment for randomization stratification factors as recorded in IXRS; Risk Difference (RD) = 5.8, 95% CI 2-sided [-3.3 to 14.9] — Risk difference (% Arm A - Arm B) based on Cochran-Mantel-Haenszel test with adjustment for randomization stratification factors as recorded in IXRS

4. Secondary Outcome: Investigator Assessed Overall Response Rate (ORR) Per IWCLL 2008 Criteria Based on Data Cutoff 03 September 2021
Description: as for outcome 3
Time Frame: Investigator assessments were done from randomization date until date of death or date of exit from study or data cut off date on 03Sep2021, whichever came first, up to 53 months of follow-up.
Population: Intent-to-treat population including all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigator's Choice
Number analyzed (Participants) | 155 | 155
Participants | 128 | 130
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigator's Choice; Test type: Other; p = 0.7340, Cochran-Mantel-Haenszel; Based on Cochran-Mantel-Haenszel test with adjustment for randomization stratification factors as recorded in IXRS; Risk Difference (RD) = -1.3, 95% CI 2-sided [-9.6 to 7.0] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was based on data cutoff date of 03Sep2021
Time Frame: From randomization date to date of death due to any cause, or date of study discontinuation, or date of data cutoff on 03Sep2021, whichever came first until 54 months of follow-up.
Population: Intent-to treat (ITT) population including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigator's Choice
Number analyzed (Participants) | 155 | 155
Months | NA [NA to NA] — Kaplan-Meier estimate for median OS and 95% CIs were not reached. | NA [NA to NA] — Kaplan-Meier estimate for median OS and 95% CIs were not reached.
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigator's Choice; Analysis stratified by factors recorded in IXRS data including presence of deletion 17 p (yes / no), ECOG (0-1/2), # of prior therapies (1-3/4+); Test type: Other; p = 0.0783, Log Rank; Log-Rank Analysis stratified by factors recorded in IXRS data: presence of deletion 17 p (yes / no), ECOG (0-1/2), # of prior therapies (1-3/4+); Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.46 to 1.04] — Cox proportional hazard analysis stratified (Arm A vs. Arm B) by factors recorded in IXRS data including presence of deletion 17 p (yes / no), ECOG (0-1/2), # of prior therapies (1-3/4+)

6. Secondary Outcome: Duration of Response (DOR) Per Independent Review Committee (IRC) Assessment Based on 15 January 2019 Data Cutoff From Interim Analysis.
Description: Duration of Response (DOR) is defined as from the first documentation of CR, CRi, PR, or nPR to the earlier of the first documentation of disease progression or death from any cause.
Time Frame: as for outcome 1
Population: Intent to treat (ITT) population including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigator's Choice
Number analyzed (Participants) | 155 | 155
Months | NA [NA to NA] — Kaplan-Meier Estimate of median DOR and 95% CI were not reached. | 13.6 [11.9 to NA] — Kaplan-Meier estimate of upper 95% CI for median DOR was not reached.
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigator's Choice; Test type: Other; p < 0.0001, Log Rank — Log Rank Test stratified by factors as recorded in IXRS, i.e., presence of del17p (Yes/No), ECOG (0-1/2), # of prior therapies (1-3/4+); Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.19 to 0.59] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Duration of Response (DOR) Per Investigator Assessment Based on 03 September 2021 Data Cutoff
Description: as for outcome 6
Time Frame: Investigator assessments were done from randomization date until date of death or study discontinuation or data cutoff date on 03Sep2021, whichever came first up to 53 months of follow-up.
Population: Intent to treat (ITT) population including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigator's Choice
Number analyzed (Participants) | 155 | 155
Months | NA [41.5 to NA] — Kaplan-Meier estimate of median DOR and upper 95% CI were not reached. | 18.3 [11.9 to 21.7]
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigator's Choice; Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.16 to 0.33] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to Next Treatment (TTNT) Based on 03 September 2021 Data Cutoff
Description: Time to Next Treatment (TTNT) is defined as the time from date of randomization to date of institution of non-protocol-specified treatment for CLL (or first dose date of acalabrutinib for Arm B subjects crossing over to receive acalabrutinib) or death due to any cause, whichever comes first.
Time Frame: From randomization date to start of non-protocol specified subsequent anticancer therapy for CLL or death due to any cause or study discontinuation or data cutoff date on 03Sep2021,, whichever came first up to 53 months of follow-up.
Population: Intent to treat (ITT) population including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Acalabrutinib Monotherapy | Arm B: Investigator's Choice
Number analyzed (Participants) | 155 | 155
Months | NA [46.9 to NA] — Kaplan-Meier estimate of median TTNT and upper 95% CI were not reached. | 22.5 [17.5 to 25.9]
Statistical Analysis 1: Comparison: Arm A: Acalabrutinib Monotherapy vs Arm B: Investigator's Choice; Test type: Other; p < 0.0001, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.21 to 0.40] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All adverse events were reported from randomization date until 30 days after the last dose of study drug or the start of new anticancer therapy (whichever comes first) up to 54 months.
Description: Data presented under All-Cause Mortality table are based on ITT Population (all randomized) as those presented in Participant Flow. Data presented under SAE and AE Tables are based on Safety Population (Subjects received at least one dose of study drug). For Arm B, adverse events are presented for Investigator's choice of IR/BR combined since the data were not reported separately for IR or BR.
Groups:
- Arm B Cross Over: Arm B Investigator Choice Crossed Over to Acalabrutinib
Arm/Group | Arm A- Acala. 100 mg BID | Arm B: Investigator Choice (IR or BR)-Main Study Period | Arm B Cross Over
All-Cause Mortality (participants affected / at risk) | 41/155 | 33/155 | 20/80
Serious Adverse Events (participants affected / at risk) | 70/154 | 86/153 | 31/80
Other Adverse Events (participants affected / at risk) | 149/154 | 145/153 | 73/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Acala. 100 mg BID (N=154) | Arm B: Investigator Choice (IR or BR)-Main Study Period (N=153) | Arm B Cross Over (N=80)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 9 (10) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Secondary immunodeficiency (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Bronchitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 3 (5) | 1 (1) | 2 (2)
Covid-19 pneumonia (Infections and infestations) | 6 (6) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 4 (4)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (14) | 13 (14) | 7 (7)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (5) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Laryngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 19 (22) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Acala. 100 mg BID (N=154) | Arm B: Investigator Choice (IR or BR)-Main Study Period (N=153) | Arm B Cross Over (N=80)
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Gastric mucosa erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0)
Gastrointestinal tract mucosal pigmentation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lip haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (16) | 24 (27) | 5 (6)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (8) | 0 (0) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 6 (7) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 9 (9) | 6 (6)
Asthenia (General disorders) | 10 (13) | 10 (13) | 6 (7)
Chest pain (General disorders) | 3 (3) | 4 (4) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (2) | 10 (10) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Extravasation (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 19 (21) | 18 (18) | 5 (5)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 5 (9) | 1 (2) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 3 (3) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 11 (12) | 8 (8) | 4 (4)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 2 (3) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 25 (33) | 29 (51) | 10 (13)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 1 (2) | 1 (1)
Swelling face (General disorders) | 1 (1) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 3 (5) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 3 (5) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 2 (3) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 2 (2) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 7 (10) | 3 (4) | 1 (1)
Immunodeficiency (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Secondary immunodeficiency (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (4) | 1 (2)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 19 (30) | 12 (14) | 3 (4)
Bronchitis pneumococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 2 (2)
Covid-19 (Infections and infestations) | 10 (10) | 4 (4) | 4 (4)
Covid-19 pneumonia (Infections and infestations) | 6 (6) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 4 (6) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 27 (52) | 17 (26) | 16 (20)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (2)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Epstein-barr virus infection reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Eye infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Hepatitis b (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 37 (75) | 67 (202) | 16 (16)
Hepatitis b reactivation (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Hepatitis c (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 6 (8) | 5 (5) | 1 (1)
Herpes zoster reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 6 (6) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 5 (5)
Nasal herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (23) | 14 (14) | 3 (3)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 3 (4) | 2 (2)
Oral fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 2 (3) | 3 (3) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 5 (5) | 2 (2) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 30 (30) | 19 (19) | 9 (9)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 5 (5) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (50) | 24 (53) | 11 (14)
Respiratory tract infection (Infections and infestations) | 18 (27) | 8 (15) | 6 (7)
Respiratory tract infection viral (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 10 (12) | 5 (6) | 1 (1)
Sinusitis (Infections and infestations) | 7 (12) | 4 (4) | 2 (2)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 31 (42) | 24 (31) | 5 (6)
Urinary tract infection (Infections and infestations) | 8 (8) | 7 (8) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 2 (3) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 13 (23) | 4 (4) | 4 (4)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eyelid contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 17 (29) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Palate injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 3 (6) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (19) | 17 (30) | 0 (0)
Aspartate aminotransferase (Investigations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 11 (11) | 4 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (23) | 13 (21) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 6 (8) | 8 (9) | 5 (5)
Blood immunoglobulin g decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urea (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Borrelia test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Candida test positive (Investigations) | 0 (0) | 2 (2) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 2 (2) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 0 (0) | 0 (0)
Faecal calprotectin increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Gamma-glutamyltransferase decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (5) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (5) | 0 (0)
Hepatitis b dna assay positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Immunoglobulins decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 10 (23) | 4 (4)
Platelet count decreased (Investigations) | 5 (12) | 6 (8) | 2 (2)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 9 (18) | 0 (0)
Weight decreased (Investigations) | 5 (6) | 6 (8) | 4 (4)
Weight increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Carbohydrate intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 6 (7) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 1 (1)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (8) | 4 (4) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 10 (11) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Vitamin k deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (24) | 8 (8) | 14 (14)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (15) | 9 (10) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (11) | 3 (4) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 2 (3) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Epstein barr virus positive mucocutaneous ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 5 (6) | 0 (0) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (14) | 2 (2) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Carotid artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 10 (17) | 3 (3) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 36 (44) | 7 (9) | 12 (14)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (12) | 8 (8) | 5 (5)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Neurosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (2)
Cytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 7 (7) | 4 (4) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulval oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvar dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (37) | 20 (29) | 8 (10)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 5 (5) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Laryngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (7) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Presbyacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (4) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (8) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 3 (3)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (8) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 15 (18) | 19 (33) | 5 (7)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (6) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (5) | 1 (1)
Accommodation disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Capillary fragility (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (4) | 0 (0)
Cataract (Eye disorders) | 4 (7) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 10 (10) | 4 (5) | 5 (5)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 11 (14) | 7 (9) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 5 (5) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 3 (3) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis superficial (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Orbital myositis (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (8) | 1 (2)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 8 (8) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8) | 5 (5) | 4 (4)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 5 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 14 (15) | 14 (14) | 2 (2)
Dental caries (Gastrointestinal disorders) | 4 (6) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 32 (45) | 64 (128) | 10 (12)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysbiosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 5 (6) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Enlarged uvula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator will not publish or publicly present any study results without prior approval or prior to 12 months following completion of the study.

DOCUMENTS (2):
  • Study Protocol (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT02970318/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT02970318/SAP_003.pdf